CLINICAL TRIAL: NCT01737112
Title: Safety and Diagnostic Performance of 99mTc-3PRGD2 SPECT/CT in Evaluation of Lung Cancer Patients
Brief Title: 99mTc-3PRGD2 SPECT/CT in Lung Cancer Patients
Acronym: TcRGDLC
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PUMCHNM05
Record Dates: First submitted 2012-11-27; First posted 2012-11-29 (Estimated); Last update posted 2017-04-07 (Actual); Status verified 2017-04

CONDITIONS: Lung Cancer
Keywords: Lung Cancer; integrin αvβ3 receptor; 99mTc-3PRGD2; SPECT/CT; efficacy and safety
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 99mTc-3PRGD2 SPECT/CT scanning (Experimental): Determine if 99mTc-3PRGD2 SPECT/CT is safe and effective in diagnosis and evaluation of lung cancer patients.
  Interventions: Drug: 99mTc-3PRGD2

INTERVENTIONS:
Drug: 99mTc-3PRGD2 — For patients in suspicion of lung cancer, single intravenous bolus injection of nearly 11.1 MBq/kg body weight of 99mTc-3PRGD2 on day one of the treatment period, whole-body planar and thoracic SPECT/CT to determine the accumulation of 99mTc-3PRGD2 in the tumors and the other parts of the body.
  Other Names: 99mTc-HYNIC-3PRGD2

SUMMARY:
This is an open-label SPECT/CT (single photon emission computed tomography / computed tomography) study to investigate the safety and diagnostic performance of 99mTc-3PRGD2 in evaluation of lung cancer patients. A single dose of nearly 11.1 MBq/kg body weight of 99mTc-3PRGD2 ( ≤ 20 µg 3PRGD2) will be intravenously injected into the patients in suspicion of lung cancer. Visual and semiquantitative method will be used to assess the whole-body planar and thoracic SPECT/CT images. Any adverse events will be collected from the patients.

DETAILED DESCRIPTION:
Integrin αvβ3 is an important member of integrin receptor family and expressed preferentially on the activated endothelial cells of angiogenesis and some types of tumor cells, but not or very low on the quiescent vessel cells and other normal cells. Therefore, the integrin αvβ3 receptor is becoming a valuable target for diagnosis and response evaluation of malignant tumors.

The tri-peptide sequence of arginine-glycine-aspartic acid (RGD) can specifically bind to the integrin αvβ3 receptor. Accordingly, a variety of radiolabeled RGD-based peptides have been developed for non-invasive imaging of integrin αvβ3 expression via single photon emission computed tomography (SPECT)or positron emission tomography (PET). Among all the RGD radiotracers studied, several RGD monomers have been investigated in clinical trials, and the preliminary results demonstrated specific imaging of various types of tumors, and the tumor uptake correlated well with the level of integrin αvβ3 expression. Recently, several RGD dimeric peptides with PEG linkers have been studied. The new types of RGD peptides showed much higher in vitro integrin αvβ3-binding affinity than the single RGD tri-peptide sequence, and importantly, they exhibited significantly increased tumor uptake and improved in vivo kinetics in animal models. As a representative, 99mTc-3PRGD2 could be easily prepared and exhibited excellent in vivo behaviors in animal models. No adverse reactions are observed in animal models to date.

For the further interests in clinical translation of 99mTc-3PRGD2, an open-label SPECT/CT study was designed to investigate the safety and diagnostic performance of 99mTc-3PRGD2 in lung cancer patients. A single dose of nearly 11.1 MBq/kg body weight 99mTc-3PRGD2 ( ≤ 20 µg 3PRGD2) will be intravenously injected into the lung cancer patients. Visual and semiquantitative method will be used to assess the whole-body planar and thoracic SPECT/CT images. Adverse events will also be observed in the patients.

ELIGIBILITY:
Inclusion Criteria:

* Males and females, ≥30 years old
* Thoracic CT and/or 18F-FDG PET/CT diagnosis in suspicion of primary or recurrent lung cancer.
* The lung cancer will be histologically confirmed or results of histology will be available.

Exclusion Criteria:

* Females planning to bear a child recently or with childbearing potential
* Known severe allergy or hypersensitivity to IV radiographic contrast.
* Inability to lie still for the entire imaging time because of cough, pain, etc.
* Inability to complete the needed examinations due to severe claustrophobia, radiation phobia, etc.
* Concurrent severe and/or uncontrolled and/or unstable other medical disease that, in the opinion of the Investigator, may significantly interfere with study compliance.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2011-02; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Visual and semiquantitative assessment of lesions and biodistribution | One year
  Visual analysis will be performed by consensus reading by at least 3 experienced nuclear medicine physician. The semiquantitative analysis will be performed by the same person for all the cases, and the tumor to background ratios(T/B) will be measured.

SECONDARY OUTCOMES:
Adverse events collection | One year
  Adverse events within 5 days after the injection and scanning of the patients will be followed and assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Fang Li, MD, Study Chair — Department of Nuclear Medicine, Peking Union Medical College Hospital, Chinese Academy of Medical Science
Locations (1):
- Department of Nuclear Medicine, Peking Union Medical College Hopital, Chinese Academy of Medical Science, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Miao W, Zheng S, Dai H, Wang F, Jin X, Zhu Z, Jia B. Comparison of 99mTc-3PRGD2 integrin receptor imaging with 99mTc-MDP bone scan in diagnosis of bone metastasis in patients with lung cancer: a multicenter study. PLoS One. 2014 Oct 22;9(10):e111221. doi: 10.1371/journal.pone.0111221. eCollection 2014. PMID 25338281